CLINICAL TRIAL: NCT02771782
Title: The Influence of BCG Vaccine as a Booster TDaP-IPV Vaccination: an Explorative Study
Brief Title: Influence of BCG on TDaP-IPV Vaccination
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BCG-DKTP1
Record Dates: First submitted 2016-02-22; First posted 2016-05-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-04

CONDITIONS: Whooping Cough
Keywords: BCG; TDaP-IPV; DPT Vaccine
MeSH Terms: conditions — Whooping Cough | interventions — BCG Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BCG (Experimental): Subjects are vaccinated with BCG vaccine (SSI) alone, 0,1ml intradermal
  Interventions: Biological: BCG vaccine (SSI)
- TDaP-IPV (Experimental): Subjects are vaccinated with TDaP-IPV vaccine (Boostrix Polio) vaccine alone, 0,5ml intramuscular
  Interventions: Biological: TDaP-IPV vaccine
- BCG+TDaP-IPV (Experimental): Subjects are vaccinated with BCG vaccine (SSI) (0.1ml intradermal) and TDaP-IPV vaccine Boostrix Polio (0.5ml intramuscular) simultaneously
  Interventions: Biological: BCG vaccine (SSI); Biological: TDaP-IPV vaccine

INTERVENTIONS:
Biological: BCG vaccine (SSI)
  Arms: BCG; BCG+TDaP-IPV
Biological: TDaP-IPV vaccine
  Arms: BCG+TDaP-IPV; TDaP-IPV

SUMMARY:
This study has three purposes:

To investigate whether the immune response to pertussis is increased when TDaP-IPV is given together with BCG vaccine, compared to when it is given alone.

To investigate whether BCG vaccination modulates the immune response to non vaccine target antigens (i.e., antigens/pathogens not used in the vaccine itself).

To investigate whether TDaP-IPV vaccination modulates the immune response to non vaccine target antigens.

DETAILED DESCRIPTION:
Rationale: The Bacillus Calmette-Guerin (BCG) vaccine not only protects against Mycobacterium tuberculosis, but has also been shown to reduce morbidity and mortality caused by non-related infections. This effect is likely due to non-specific immunomodulatory effects, at least in part on the innate immune system. Additionally, BCG has been shown to improve immunogenicity of other vaccinations. In contrast, whilst the diphtheria-tetanus-pertussis (DTP) combination vaccine protects against infection with Bordetella pertussis, Clostridium tetani and Corynebacterium diphtheria, it has also been associated with increased mortality due to unrelated infections, particularly in girls in high-mortality countries.

Although widespread DTP vaccination has initially reduced pertussis mortality, the disease has persisted and recently resurged in a number of countries with highly vaccinated populations, including the Netherlands. This has been partially attributed to the switch from a whole-cell vaccine (which is still being used in low-income countries) to a more defined acellular pertussis vaccine, which only protects for a limited period (5-8 years). Strategies to improve the efficacy of pertussis vaccination are therefore urgently required.

As the BCG vaccine has already been used to improve the immunogenicity of other vaccines, the investigators hypothesize that BCG vaccination before or at the same time of DTP vaccination increases the immunogenicity of the DTP vaccine in terms of antibody and T-cell responses to pertussis. Moreover, the investigators aim to assess the effect of DTP vaccination on the known long-term beneficial non-specific effects of BCG on non-mycobacterial infections.

Objective: To examine the effect of BCG as an adjuvant on DTP vaccination, and to investigate the non-specific training effects of BCG and DTP, alone and in combination, on the innate immune system.

Study population: Healthy adult volunteers.

Main study parameters: Comparison of pertussis-specific antibody and T-cell responses, as well as gene transcription between BCG, TDaP-IPV and BCG+TDaP-IPV vaccinated groups. Comparison of cytokine responses to unrelated antigens and/or pathogens before and after BCG, TDaP-IPV or BCG+TDaP-IPV vaccination.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no direct benefit to the study participants but these results will potentially lead to novel strategies to optimize vaccinations. The risks for participants are negligible, with the only expected risks being minor side-effects from vaccination and local hematoma forming at the site of venepuncture. This will be minimized by the performance of these procedures by experienced personnel.

ELIGIBILITY:
Inclusion Criteria:

* healthy females

Exclusion Criteria:

* systemic medication use other than oral contraceptive drugs
* history of disease resulting in immunodeficiency
* previous vaccination with BCG
* pregnancy
* allergy to neomycin or polymyxin
* known previous allergic reaction to vaccination with diphteria, tetanus, pertussis or polio vaccines
* One of following phenomena after previous vaccination with pertussis containing antigens: Fever >40 °C within 48 hours after vaccination, hypotonous-hyporesponsiveness episode within 48 hours after vaccination, convulsions with or without fever within 3 days after vaccination

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Antibody response to TDaP-IPV | 2 weeks
  antibody titers to antigens in the TDaP-IPV (PT, FHA, Prn, DT, TT) will be measured.
Antibody response to TDaP-IPV | 3 months
  antibody titers to antigens in the TDaP-IPV (PT, FHA, Prn, DT, TT) will be measured.
Antibody response to TDaP-IPV | 1 year
  antibody titers to antigens in the TDaP-IPV (PT, FHA, Prn, DT, TT) will be measured.
T-cell response to TDaP-IPV | 2 weeks
  T-cell responses will be measured by FACS
T-cell response to TDaP-IPV | 3 months
  T-cell responses will be measured by FACS
T-cell response to TDaP-IPV | 1 year
  T-cell responses will be measured by FACS
PBMC cytokine response to pertussis related antigens | 2 weeks
  IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g
PBMC cytokine response to pertussis related antigens | 3 months
  IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g
PBMC cytokine response to pertussis related antigens | 1 year
  IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g
B-cell phenotype analysis | 2 weeks
  pertussis specific B-cells will be analyzed by FACS
B-cell phenotype analysis | 3 months
  pertussis specific B-cells will be analyzed by FACS
B-cell phenotype analysis | 1 year
  pertussis specific B-cells will be analyzed by FACS

SECONDARY OUTCOMES:
PBMC responses to heterologous antigens | 1 day
  PBMCs will be stimulated with LPS, S. aureus, C.albicans, PHA, S.pneumoniae, zymosan. Responses on cytokine levels (IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g) and ROS production will be measured
PBMC responses to heterologous antigens | 4 days
  PBMCs will be stimulated with LPS, S. aureus, C.albicans, PHA, S.pneumoniae, zymosan. Responses on cytokine levels (IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g) and ROS production will be measured
PBMC responses to heterologous antigens | 2 weeks
  PBMCs will be stimulated with LPS, S. aureus, C.albicans, PHA, S.pneumoniae, zymosan. Responses on cytokine levels (IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g) and ROS production will be measured
PBMC responses to heterologous antigens | 3 months
  PBMCs will be stimulated with LPS, S. aureus, C.albicans, PHA, S.pneumoniae, zymosan. Responses on cytokine levels (IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g) and ROS production will be measured
PBMC responses to heterologous antigens | 1 year
  PBMCs will be stimulated with LPS, S. aureus, C.albicans, PHA, S.pneumoniae, zymosan. Responses on cytokine levels (IL-6, TNF, IL-1b, IL-10, IL-17, IL-22, IFN-g) and ROS production will be measured
Transcriptional profile of PBMCs | 1 day
  Transcriptional profile of PBMCs will be measured by RNAseq to assess for active gene transcription programs
Transcriptional profile of PBMCs | 4 days
  Transcriptional profile of PBMCs will be measured by RNAseq to assess for active gene transcription programs
Transcriptional profile of PBMCs | 2 weeks
  Transcriptional profile of PBMCs will be measured by RNAseq to assess for active gene transcription programs
Transcriptional profile of PBMCs | 3 months
  Transcriptional profile of PBMCs will be measured by RNAseq to assess for active gene transcription programs
Epigenetic markers of monocytes | 1 day
  Levels of activating and inhibiting epigenetic marks will be assessed
Epigenetic markers of monocytes | 4 days
  Levels of activating and inhibiting epigenetic marks will be assessed
Epigenetic markers of monocytes | 2 weeks
  Levels of activating and inhibiting epigenetic marks will be assessed
Epigenetic markers of monocytes | 3 months
  Levels of activating and inhibiting epigenetic marks will be assessed

OTHER OUTCOMES:
Leukocyte differential count | 1 day,
  Leukocyte differential counts will be performed
Leukocyte differential count | 4 days
  Leukocyte differential counts will be performed
Leukocyte differential count | 2 weeks
  CBC parameters will be measured before and after vaccination
Leukocyte differential count | 3 months
  Leukocyte differential counts will be performed
Leukocyte differential count | 1 year
  Leukocyte differential counts will be performed
NK cell phenotype | 2 weeks
  NK cell activation markers will be assessed by FACS
NK Cell phenotype | 3 months
  NK cell activation markers will be assessed by FACS
NK cell phenotype | 1 year
  NK cell activation markers will be assessed by FACS
NK cell function | 2 weeks
  degranulation of NK cells upon stimulation with tumor cells will be assessed
NK cell function | 3 months
  degranulation of NK cells upon stimulation with tumor cells will be assessed
NK cell function | 1 year
  degranulation of NK cells upon stimulation with tumor cells will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Netea, Prof. Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Radbdoudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blok BA, de Bree LCJ, Diavatopoulos DA, Langereis JD, Joosten LAB, Aaby P, van Crevel R, Benn CS, Netea MG. Interacting, Nonspecific, Immunological Effects of Bacille Calmette-Guerin and Tetanus-diphtheria-pertussis Inactivated Polio Vaccinations: An Explorative, Randomized Trial. Clin Infect Dis. 2020 Jan 16;70(3):455-463. doi: 10.1093/cid/ciz246. PMID 30919883